CLINICAL TRIAL: NCT04970589
Title: Enhancing Efficacy of Mango Phytochemicals in Cognitive Function and Cardiometabolic Health in Lean and Obese
Brief Title: Enhancing Efficacy of Mango Polyphenols in Lean and Obese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Susanne Talcott, PhD, Assoc. Professor, Texas A&M University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TexasAMU-IRB2018-0405F
Record Dates: First submitted 2021-07-06; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Mangifera indica extract; Probiotics

STUDY DESIGN:
Intervention Model Description: Group 1: BMI 18-23: 400g of mango and a placebo capsule every day for 8 weeks Group 2: BMI 18-23: 400g of mango and a probiotic capsule every day for 8 weeks Group 3: BMI 27-35: 400g of mango and a placebo capsule every day for 8 weeks Group 4: BMI 27-35: 400g of mango and a probiotic capsule every day for 8 weeks
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lean/Placebo Capsule (Placebo Comparator): Participants (Lean:BMI 18-23) will be asked to take 400g of mango and a placebo capsule every day for 8 weeks
  Interventions: Other: Mango; Other: Placebo
- Lean/Probiotics (Experimental): Participants (Lean:BMI 18-23) will be asked to take 400g of mango and a probiotic capsule every day for 8 weeks
  Interventions: Other: Mango; Dietary Supplement: Probiotics
- Obese/Placebo Capsule (Experimental): Participants (Obese:BMI 27-35) will be asked to take 400g of mango and a placebo capsule every day for 8 weeks
  Interventions: Other: Mango; Other: Placebo
- Obese/Probiotics (Experimental): Participants (Obese:BMI 27-35) will be asked to take 400g of mango and a probiotic capsule every day for 8 weeks
  Interventions: Other: Mango; Dietary Supplement: Probiotics

INTERVENTIONS:
Other: Mango — 400g of mango/day
Dietary Supplement: Probiotics — 1 probiotics capsule/day
  Arms: Lean/Probiotics; Obese/Probiotics
Other: Placebo — 1 Placebo capsule/day
  Arms: Lean/Placebo Capsule; Obese/Placebo Capsule

SUMMARY:
The objective of this research is to determine beneficial impact of mango phytochemicals in lean and obese individuals for cognitive function and gut health. Investigate how obesity impacts the efficacy of mango polyphenols on cognitive function and health. Investigate the ability of probiotic bacteria to optimize the absorption and efficacy of mango phytochemicals in lean and obese individuals.

DETAILED DESCRIPTION:
Rationale: In obesity, interactions between adipocytes and macrophages are of increasing importance to understanding obesity and chronic diseases. Dietary compounds, such as polyphenols, are expected to cause significant changes in inflammatory biomarkers in lipid tissue that are different from those in blood. To capture any changes of macrophages interacting with lipid tissue and associated biomarkers, lipid biopsies were collected in this study.

Before the study day: Participants were advised to not eat anything after dinner at 7-8pm the night (A 12-hour fast). Drink plenty of water, at least 8 fl oz in the evening and 8 fl oz in the morning. Participants were advised to eat a well-balanced meal consisting of 25% protein-rich food, 25% whole grain high-fiber carbohydrate, and 50% fruits and vegetables prior to beginning of fast. Prior to the first study session, participants were asked to fill out a 72-h nutritional report with all food and drinks consumed using a website (www.mynetdiary.com)

Study day: Participants were asked to consume 400 g of cubed, fresh mango during the early morning hours of the study day starting right after the baseline blood draw. If they were in the placebo group, they were asked to take one placebo capsule daily. The placebo used in this study consisted of vegetable cellulose (HPMC USP) filled with 100% microcrystalline cellulose USP. If they were in the probiotic group, they were asked to take one capsule of the Renew Life Ultimate Flora "Extra Care" probiotic daily.

Study Treatment: In this study participants were placed into one of four different groups depending on their BMI. The study treatment depended on which study group they were in:

BMI 18-23, Group 1: They were asked to consume a single portion of 400g of mango and take one placebo capsule every day for the duration of the 8-week study.

BMI 18-23, Group 2: They were asked to consume a single portion of 400g of mango and take one probiotic capsule every day for the duration of the 8-week study.

BMI 27-35, Group 1: They were asked to consume a single portion of 400g of mango and take one placebo capsule every day for the duration of the 8-week study.

BMI 27-35, Group 2: They were asked to consume a single portion of 400g of mango and take one probiotic capsule every day for the duration of the 8-week study.

Subjects did not know if they received probiotic or placebo capsules as part of their study treatment. During all sessions, subjects were asked questions about their general health.

Study Session 1 (Days 1-3): Blood samples (30 mL or 6 teaspoons each) were taken before and 2 hours after mango consumption (Days 1, 2, and 3) by the study phlebotomist. Subjects were asked to collect approximately 3 fl. oz (half a cup) of urine in the morning of Days 1, 2, and 3, and 3 fl. ox (half a cup) in the evening of Days 1 and 2. They were also asked to collect a stool sample to bring on Day 1. The researchers gave the subjects containers for the urine and a kit for stool collection, as well as instructions on how to collect each of those samples. Instructions on how to transport those samples were also given to them. During Study Session 1 (Day 1), subjects took two cognitive function tests (Trail Making and Digit Span).

Study Session 2 (Day 29): The study phlebotomist collected a single blood sample (30 mL or 6 teaspoons) from the subject's arm. Participants were also asked to collect a stool sample using a collection kit we will provide.

NeuroTracker Sessions: During the last two weeks of the study (between days 43 and 56), subjects were asked to come to our facility to perform a total of ten sessions using the NeuroTracker, a cognitive function test. They could perform up to one session per day, and all ten sessions were completed between days 43 and 56. Before each session, subjects were asked to fill out the NeuroTracker questionnaire (to assess their emotional, mental, and physical state) and a food log.

Study Session 3 (Days 54-56): Blood samples (30 mL or 6 teaspoons each) were taken right before and 2 hours after mango consumption (Days 54, 55, and 56) by the study phlebotomist. Subjects were asked to collect approximately 3 fl. oz (half a cup) of urine in the morning of Days 54, 55, and 56, and 3 fl. ox (half a cup) in the evening of Days 54 and 55. They were also asked to collect a stool sample to bring on Day 54. The researchers gave the subjects containers for the urine and a kit for stool collection, as well as instructions on how to collect each of those samples. Instructions on how to transport those samples were also given to them. During this session (Day 54), subjects took two cognitive function tests (Trail Making and Digit Span). On Day 56, we measured the participant's body fat using an Omron Handheld Body Fat Monitor.

Cognitive Function Testing: On Days 1 and 54, we assessed the cognitive function of the subjects by giving them the following tests: The Trail Making Test (TMT A&B) and the Wechsler Adult Scale-Revised Digit Span test.

During the last two weeks of the study (between days 43 and 56), subjects were also run through our NeuroTracker program. This was to test their spatial awareness. The TMT A&B Test assesses measure of attention, speed, mental flexibility, spatial organization, visual pursuits, recall, and recognition. The Wechsler Adult Scale-Revised Digit Span is a measure of mental tracking, memory, and mental flexibility.

Lipid biopsy - Optional: This study included an optional lipid biopsy component and participants were free to agree to participate in this procedure at the beginning and end of this study.

This procedure was performed under supervision of the study physician Dr. Bramhal and performed by Dr. Jim Fluckey and Dr. Steven Riechman.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* BMI between 18-23 and 27-35

Exclusion Criteria:

* History of acute cardiac event, stroke, or cancer
* Alcohol or substance abuse within the last 6 months
* Pregnancy or lactation (or planned pregnancy)
* No recurrent hospitalizations within the last 6 months
* Allergy against any of the study treatments (mango or probiotics)
* Liver or renal dysfunction
* Hepatitis B or C, HIV
* Currently smoking more than 1 pack/week
* History of dizziness/fainting during/after blood draws

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Cognitive Function (NeuroTracker) | From Week 6 to Week 8
  NeuroTracker: Ten sessions should be completed between days 43 and 56. Fill out the NeuroTracker questionnaire to assess their emotional, mental, and physical state.
Cognitive Function (The Trail Making Test) | At baseline and week 8
  The Trail Making Test (TMT A&B) On Days 1 and 54, Assessed the cognitive function of the subjects by giving them these tests. The TMT A&B Test assesses measure of attention, speed, mental flexibility, spatial organization, visual pursuits, recall, and recognition.
Cognitive Function (the Wechsler Adult Scale-Revised Digit Span test) | At baseline and week 8
  The Wechsler Adult Scale-Revised Digit Span test: On Days 1 and 54, Assessed the cognitive function of the subjects by giving them these tests. The Wechsler Adult Scale-Revised Digit Span is a measure of mental tracking, memory, and mental flexibility.

SECONDARY OUTCOMES:
Changes from baseline in the levels of Inflammatory biomarkers in plasma | At baseline and week 8
  Measure the Inflammatory biomarkers including TNF-a, IL-1b, IL-6, IL-8, IL-10.
Change from baseline in the levels of metabolites of gallic acid in urine and plasma after mango intake. | At baseline and week 8
  Aliquoted urine and plasma samples were thawed and centrifuged at 13,000 x g for 10 mins at 4°C immediately prior to analysis by HPLC-MSn. All quantification of metabolites (pyrogalloyl-O-glucuronide, O-methyl-gallic acid, O-methylgallic acid-O-sulfate, O-methylpyrogalloyl-O-sulfate, pyrogalloyl-O-sulfate, deoxypyrogallol-O-sulfate, O-methylpyrogalloyl-O-sulfate) was performed in full MS and expressed as gallic acid equivalents.
Change from baseline in gut microbiota composition in stool samples | At baseline and week 8
  16S rRNA-based pyrosequencing to quantify bacterial taxa

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Talcott, Ph.D, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States